CLINICAL TRIAL: NCT06275256
Title: Outcomes of Minimally Invasive Surgical Treatments (MIST) for Benign Prostatic Hyperplasia (BPH): A Single-Institution Prospective Study
Brief Title: Outcomes of MIST for BPH: A Single-Institution Prospective Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Premal Patel, MD, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS26226
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Rezum (Experimental): This arm will receive the Rezum procedure.
  Interventions: Procedure: Rezum
- iTind (Experimental): This arm will receive the iTind Procedure
  Interventions: Device: iTind

INTERVENTIONS:
Procedure: Rezum — The Rezum device is inserted, a needle is deployed, and vapor is injected into the prostate for nine seconds. This vapor disperses between cells, then cools, releases heat, and gently disrupts the prostate's cells. Because of the initial swelling, a catheter is then inserted, which will remain for two to five days.
  Arms: Rezum
Device: iTind — The iTind device is temporarily placed inside the prostatic urethra (the narrowed portion of the prostate), where it slowly expands and exerts gentle pressure at three precise points. The effect of the iTind is to widen the prostatic urethral opening through which urine can now flow more easily.
  Arms: iTind

SUMMARY:
The investigators wish to perform a prospective study at the Men's Health Clinic in Winnipeg, Manitoba to accomplish two goals: 1) Prospectively describe 1 year outcomes for MIST therapies performed at the clinic 2) perform a head to head comparison of Rezum water vapor therapy vs the iTind device in respect to symptom score improvement, uroflow parameters and side effect profile.

DETAILED DESCRIPTION:
This prospective study is to be conducted at the Men's Health Clinic in Winnipeg, Manitoba. All eligible patients who are to undergo Rezum or iTind procedure for BPH/LUTS between March 2024 and March 2025 are to be included in the study. Patient meeting inclusion criteria and exclusion criteria will be recruited to participate in this study.

Inclusion criteria: patients > 18 years of age, undergoing Rezum or iTind treatment Exclusion criteria: ASA III or higher, active UTI within past week, age < 18 years of age, no informed consent Follow-up/data measurements will occur pre-procedure, immediately post procedure, 1 week, 6 weeks, and 3 months following procedure. At time of consultation pre-procedure, baseline symptom scores, uroflow parameters will be obtained. VAS pain score is to be obtained during procedure, immediately post procedure, and at time of catheter or device removal 1 week post procedure. Uroflow parameters and symptoms scores will be again measured at 6 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years of age undergoing Rezum or iTind treatment

Exclusion Criteria:

* ASA 3 or higher, active UTI within past week, age < 18 years of age, no informed consent

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Symptom Scores | 1, 3, 6 months post-procedure
  Using the IPSS (International Prostate Symptom Score) questionnaires to measure improvement in symptom scores
Uroflow | 1, 3, 6 months post-procedure
  Measuring uroflow parameters such as Qmax pre and post procedure
Uroflow | 1, 3, 6 months post-procedure
  Measuring uroflow parameters such as PVR (post-void residual volume) pre and post procedure
Symptom Scores | 1, 3, 6 months post-procedure
  Using the MHSQ-EjD (Male Sexual Health Questionnaire) questionnaire to measure changes in symptom scores
Symptom Scores | 1, 3, 6 months post-procedure
  Using the IIEF-15 (Index of Erectile Function) questionnaire to measure changes in symptom scores
Symptom Scores | 1, 3, 6 months post-procedure
  Using the OAB-qSF (overactive bladder symptom and health-related quality of life short-form questionnaire) to measure changes in symptom scores

SECONDARY OUTCOMES:
Pain Scale | 1, 3, 6 months post-procedure
  Using a visual analogue pain scale [range 0-10; 0 = no pain, 10 = maximal pain], pain will be assessed as reported by the patient post-operatively to determine their pain

CONTACTS AND LOCATIONS:
Locations (1):
- Men's Health Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No